CLINICAL TRIAL: NCT02057809
Title: Investigation of "Family-centered" Pediatric Rehabilitation Services Received by Children With Developmental Disabilities
Brief Title: "Family-centered" Pediatric Rehabilitation Services in Children With Developmental Disabilities
Status: Completed | Type: Observational
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Lin-Ju Kang, Assistant Professor, Chang Gung University
Other Study IDs: 102-3767B
Record Dates: First submitted 2013-12-22; First posted 2014-02-07 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Developmental Disabilities; Autistic Spectrum Disorder
Keywords: Developmental Disabilities; Family-centered services; Pediatric rehabilitation
MeSH Terms: conditions — Developmental Disabilities; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Parent-child dyad: Children with Developmental Disabilities and their parents
- Therapits: Therapists experienced in serving children with developmental disabilities

SUMMARY:
Developmental disability is a severe chronic disabled condition caused by mental or physical impairments. Children with developmental disabilities may face life-long difficulties in motor functioning, self-care, condition, communication, and independent living. They often receive rehabilitation services to promote daily functions and participation in home, school, and community lives.

"Family-centered" service has been considered as "best practice" in pediatric rehabilitation. Therapists encourage children with developmental disabilities and their parents to participate in decision making and implementing process of intervention, and provide intervention plan that best fit their family needs. Research shows that for children with developmental disabilities, family-centered services can enhance children's development, decrease parenting stress, promote emotional wellness, and increase parental satisfaction to services. Though the "family-centered" concept has been considered as relevant in pediatric rehabilitation, there are still difficulties, as well as a lack of evidence regarding its implementation in practice.

Reflecting the trend of family-centered medical care, the benefits of national health insurance in Taiwan for early intervention outpatient care will emphasize on family-centered intervention. The range of benefits may include communication with parents, parental education, consultation and instructions for home programs. Besides, outcomes of family-centered intervention will be treated as an important index for monitoring the quality of medical services.

Given that there is a lack of investigation regarding the family-centered pediatric rehabilitation, the purposes of this one-year research project are to investigate the implementation of family-centered pediatric rehabilitation for children with developmental disabilities and to identify related influencing factors. This study will provide empirical evidence for family-centered services in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. children aged 2 to 12 years.
2. children with a primary diagnose or condition associated with developmental disabilities, including attention deficit hyperactivity disorder, autism, intellectual disability, Down syndrome, learning disorders, cerebral palsy, and other developmental delay.
3. parents agree to participate in this study.

Exclusion Criteria:

1. children with unstable physical conditions, such as cancer, having surgery within 3 months, infection, or other active medical conditions.
2. children with progressive disease (e.g. neuromuscular disease) or degenerative disorders (e.g. degenerative seizures).

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with developmental disabilities (DD) aged 2-12 years. Children with DD refer to a diverse group of severe, chronic disability that is attributed to mental and/or physical impairments, resulting in substantial functional limitations in major life activity.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The Measure of Processes of Care-20 | 1 year

SECONDARY OUTCOMES:
Measure of Processes of Care- for Service Providers | 1 year
Children and Adolescent Factor Inventory | 1 year
Assessment of Preschool Children's Participation (APCP) | 1 year
Children's Assessment of Participation and Enjoyment (CAPE) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Ju Kang, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan